CLINICAL TRIAL: NCT02841254
Title: Diagnostic Performance of Clinical Signs Patients Suspected of Meningitis to Emergencies. Prospective and Multicentric Study
Brief Title: Diagnostic Performance of Clinical Signs Patients Suspected of Meningitis to Emergencies
Acronym: MEDWATCH
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_0102
Record Dates: First submitted 2016-07-19; First posted 2016-07-22 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Meningitis
MeSH Terms: conditions — Meningitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Non interventional study

SUMMARY:
Meningitis are serious infections. Evidenced by high rates of mortality and sequelae. However, these diseases have a relatively small impact. Also physician services Home Emergencies they must be vigilant, alert, for clinical signs to be suspected meningitis. Indeed, it is only after this essential clinical milestone that will be carried out a lumbar puncture which will confirm the diagnosis and to quickly begin treatment.

Unfortunately, if recent studies can improve the therapeutic management of patients with meningitis, no study was interested in yet fundamental step of diagnosis.

It seems therefore necessary to achieve a prospective clinical study to reassess the adequacy of the clinical signs in the diagnosis of meningitis. The ideal would be to achieve a predictive clinical score of the presence or absence of meningitis.

ELIGIBILITY:
Inclusion Criteria:

May be included in the study two groups of patients:

*On the one hand, those in which will be carried out a lumbar puncture. Ideally, all patients in whom the examination is envisaged will be included. The logistics must allow inclusion rate as high as possible (see below).

So, are included in this group, patients for which the following criteria are met:

* Over 15 years patient and 3 months,
* Admission to the emergency for less than 6 hours
* Realization of a proposed lumbar puncture,
* Information sheet given. *On the other hand, those in whom it is not intended to be carried by lumbar puncture, but for which the clinical picture present on admission makes relevant for clinical signs of meningitis.

So, are included in this group, patients for which the following criteria are met:

* Over 15 years patient and 3 months,
* Admission to the emergency for less than 6 hours
* At least one of the following 5 clinical signs motivating consultation and / or present on admission:

  * fever (measured temperature above 38 ° C)
  * headache,
  * vomiting,
  * stiff neck,
  * vigilance disorders,
* Information sheet given.

Exclusion Criteria:

* Patient who underwent neurosurgery recent (within the month before admission).

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients visiting the Adults Emergency
Sampling Method: Non-Probability Sample
Enrollment: 579 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
meningitis (either viral or bacterial) or absence of meningitis | Until 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Cédric BRETONNIERE, Dr, Principal Investigator — Nantes University Hospital
Locations (3):
- France (3):
  - Châteaubriant Hospital, Châteaubriant
  - Nantes University Hospital, Nantes
  - Saint-nazaire Hospital, Saint-Nazaire

IPD SHARING:
Plan to Share IPD: No